CLINICAL TRIAL: NCT00221468
Title: A Single-Blind Prospective Study of Quetiapine for the Treatment of Mood Disorders in Adolescents
Brief Title: A Study of Quetiapine for the Treatment of Mood Disorders in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRUSQUET0296
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2007-03

CONDITIONS: Mood Disorders
Keywords: Adolescents
MeSH Terms: conditions — Mood Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Quetiapine (Experimental): Patients will begin 100mg of quetiapine on day 1 and titrated to a maximum dose of 400mg by day 4, with flexible dosing to 600mg by day 28. The total duration of treatment will be 84 days (12 weeks).
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: quetiapine — 100mg of quetiapine on day 1 and titrated to a maximum dose of 400mg by day 4, with flexible dosing to 600mg by day 28. The total duration of treatment will be 84 days (12 weeks).
  Other Names: Seroquel

SUMMARY:
The purpose of this research study is to obtain preliminary data regarding the effectiveness, tolerability, and safety of quetiapine therapy for adolescents who have a mood disorder and have at least one parent with bipolar disorder (severe mood swings).

DETAILED DESCRIPTION:
Bipolar disorder is a common, life-long, progressive disease that typically begins in adolescence or early adulthood and is associated with significant morbidity and mortality (Lish et al., 1994). Family studies have shown that offspring of parents with bipolar disorder have a 30% chance of developing a mood disorder, while children with both parents with a mood disorder (with at least one with bipolar disorder) have a 70% chance of developing a mood disorder (Goodwin and Jamison 1990). Indeed, children (< 18 years old) have an even greater risk for developing bipolar disorder if they have a parent with the disorder (reviewed in Lapalme et al., 1997; DelBello and Geller, 2002; Chang and Steiner, 2003). Since the clinical manifestations of bipolar disorder often present early in life and may worsen with age, it is imperative that this illness is recognized and treated as readily as possible. Bipolar disorder may have a number of prodromal or early-onset presentations that do not include syndromal mania. These prodromes may include cyclothymia, dysthymia, and subsyndromal manic, depressive, and mixed affective symptoms (Chang et al., 2000, reviewed in Lapalme et al., 1997).

There have been several investigations of divalproex for the treatment of mood symptoms in children at familial risk for bipolar disorder (Chang et al., 2002; Findling et al., 2002). Chang et al., found a significant reduction in mood symptoms and improvement in overall functioning following treatment with divalproex in 23 children who did not have bipolar I disorder but who were diagnosed with mood symptoms/syndromes and who had a parent with bipolar disorder (Chang et al., 2002). Similarly, Findling et al. reported that children with mood symptoms and a multigenerational family history of bipolar disorder had a significant reduction in mood symptoms when treated with divalproex compared with placebo (Findling et al., 2002). To our knowledge, there have been no studies evaluating the use of atypical antipsychotics for the treatment of children at familial risk for developing bipolar disorder who are diagnosed with mood disorders other than bipolar I disorder.

Controlled investigations suggest that quetiapine is effective for the treatment of mania in adults and adolescents (Adityanjee and Schulz, 2003; Sachs et al., 2002; DelBello et al., 2002). Additionally, quetiapine is particularly well-tolerated and safe in children and adolescents (DelBello et al., 2002; Findling, 2003). Our group has reported that children at risk for bipolar disorder exhibit neurochemical abnormalities, suggesting neuronal damage may occur prior to the onset or early in the course of a mood disorder. Furthermore, recent laboratory studies suggest that quetiapine may have neuroprotective properties (Xu et al., 2002). Therefore, quetiapine is the ideal choice for the treatment of adolescents at familial risk for developing bipolar disorder who are presently exhibiting a mood disorder.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, subjects must meet the following criteria:

1. Male or female patients, 12-18 years of age.
2. Female patients of menarche must be using a medically accepted means of contraception (e.g. oral contraceptives, Depo-Provera, abstinence).
3. Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent. Each patient must also give assent to study participation.
4. Patients must have a diagnosis of a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) mood disorder (dysthymia, major depressive disorder, depressive disorder not otherwise specified, cyclothymic, bipolar I disorder, bipolar II disorder, or bipolar disorder not otherwise specified) as determined by the Washington University at St. Louis Kiddie Schedule of Affective Disorders and Schizophrenia (WASH-U K-SADS) (Geller et al., 2000).
5. Patients must currently display symptoms of depression/dysthymia (Childhood Depression Rating Scale > 35) or mania/hypomania (Young Mania Rating Scale > 14).

Exclusion Criteria:

Patients will be excluded from the protocol for any of the following reasons:

1. Female patients who are either pregnant or lactating.
2. Clinically significant or unstable hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, hematologic, or other systemic medical conditions.
3. Neurologic disorders including epilepsy, stroke, or severe head trauma.
4. Clinically significant laboratory abnormalities on any of the following tests: complete blood count (CBC) with differential, electrolytes, BUN, creatinine, hepatic transaminases, thyroid stimulating hormone (TSH), and electrocardiogram (EKG).
5. Mood symptoms due to a general medical condition or substance-induced mania (DSM-IV).
6. Mental retardation (intelligence quotient [IQ] < 70).
7. History of hypersensitivity to or intolerance to quetiapine.
8. Prior history of quetiapine non-response.
9. DSM-IV substance (except nicotine or caffeine) dependence within the past 3 months.
10. Judged clinically to be at serious suicidal risk.
11. Participation in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry.
12. Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections and day 0.
13. Treatment with concurrent mood stabilizers or anticonvulsants, benzodiazepines (except as described below), psychostimulants, guanethidine, or guanadrel, or antidepressants.
14. Schizophrenia or other psychotic disorders (including schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, or psychotic disorder not otherwise specified) as defined in the DSM-IV.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2003-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Improvement (CGI) | 12 weeks
  The Clinical Global Impression Improvement Score of < 2 (much or very much improved) will be used to quantify the adolescent's change in overall severity of illness.

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) | 12 weeks
  The Young Mania Rating Scale (YMRS) will be used as a measure of efficacy (change in YMRS total scores from baseline to endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States